CLINICAL TRIAL: NCT07233200
Title: Serial Dermabrasion for Aesthetic Enhancement of Free Flap Skin Paddles and Donor Sites: A Prospective Split-Flap/Scar Controlled Study
Brief Title: Dermabrasion for Free Flap Aesthetic Enhancement
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Jessyka Lighthall, Chief, Facial Plastic and Reconstructive Surgery, Professor, Department of Otolaryngology-Head and Neck Surgery, Milton S. Hershey Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00027645
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Scar Conditions and Fibrosis of Skin
Keywords: scar; head and neck reconstruction; dermabrasion; aesthetics
MeSH Terms: conditions — Cicatrix | interventions — Dermabrasion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Split scar (Experimental): Free flap scars will be split and half treated, half untreated for comparison
  Interventions: Device: Dermabrasion

INTERVENTIONS:
Device: Dermabrasion — This is the only intervention. Free flap scars will be split and half treated, half untreated then outcomes graded.

SUMMARY:
The purpose of this study is to evaluate the aesthetic benefit and safety of serial dermabrasion for free flap skin paddles and donor site scars in head and neck reconstruction.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18 years or older.
2. History of successful free flap reconstruction with a cutaneous skin paddle in the head and neck region.
3. Patients with benign (eg. osteoradionecrosis, trauma) or malignant (eg. squamous cell carcinoma) diagnoses requiring free flap reconstruction.
4. Benign free flap patients must be a minimum 3 months post-operative to ensure flap maturity. Malignant free flap patients must be a minimum of 3 months post-operative or post-radiation with no further cancer treatment (eg. radiation, surgery, chemotherapy) planned at that time.
5. Flap skin paddle must be of sufficient size and external to allow for split-treatment design (minimum 4 cm in diameter). Donor site scar must also be sufficient size (minimum 6 cm in length)
6. Patients must have ability to provide informed consent.
7. Willingness and ability to comply with the treatment and follow-up schedule.

Exclusion Criteria:

1. Inability to give informed consent.
2. Evidence of active flap or radiation skin complications (e.g., infection, partial necrosis, wound breakdown).
3. Completion of head and neck radiation therapy within 3 months of first dermabrasion treatment date.
4. Uncontrolled diabetes mellitus (HbA1c > 8.0%).
5. Current antibiotic use or known immunocompromised state.
6. History of keloid formation or hypertrophic scarring.
7. Fitzpatrick skin type VI or higher (due to increased risk of pigmentary changes).
8. Use of isotretinoin medication within the past 3 month (known to induce photosensitivity).
9. Current use of blood thinners that cannot be safely paused.
10. Known photosensitivity disorders.
11. Active malignancy requiring ongoing treatment.
12. Inability or unwillingness to avoid sun exposure during the treatment period.
13. Inability to perform or adhere to prescribed wound care.
14. Inability or unwillingness to attend follow-up visits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-07-01 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Aesthetic grading of treated area compared to untreated | 1, 3, and 6 months post-treatment
  Aesthetic improvement of the treated half of the free flap skin paddle/donor site scar, as compared to the untreated half. This will be measured through blinded evaluations of standardized clinical photographs. Each side of the skin paddle or donor site scar will be labeled as side 1 or 2.

CONTACTS AND LOCATIONS:
Overall Officials: Jessyka G Lighthall, Principal Investigator — Milton S. Hershey Medical Center

IPD SHARING:
Plan to Share IPD: No